CLINICAL TRIAL: NCT01925885
Title: Focal Impulse and Rotor Modulation Ablation Trial for Treatment of Paroxysmal Atrial Fibrillation (FIRMAT-PAF)
Acronym: FIRMAT-PAF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: •Terminated: recruiting or enrolling participants has halted prematurely and will not resume; participants are no longer being examined or treated
Sponsor: Indiana University (Other)
Collaborators: University of California, Los Angeles (Other); Topera, Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IU-1302010649
Record Dates: First submitted 2013-08-05; First posted 2013-08-20 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PVI Ablation (Active Comparator): Standard of care arm-pulmonary vein isolation (PVI)-involving moving the ablation catheter from point to point in a continuous line to surround the the orifices of the pulmonary veins in order to eliminate electrical conduction between the veins and left atrium.
  Interventions: Procedure: PVI Ablation
- FIRM Ablation (Experimental): FIRM ablation for paroxysmal atrial fibrillation at sites of rotors or focal impulse formation as designated by using the mapping algorithm of RhythmView
  Interventions: Procedure: FIRM Ablation

INTERVENTIONS:
Procedure: PVI Ablation — PVI ablation for atrial fibrillation specifically targets areas in the left atrium in the area just outside the pulmonary veins to eliminate triggers of atrial fibrillation.
  Other Names: Ablation; Atrial Fibrillation; Arrhythmia; Radiofrequency Ablation; Mapping; Pulmonary Veins; Paroxysmal Atrial Fibrillation
  Arms: PVI Ablation
Procedure: FIRM Ablation — Ablation for atrial fibrillation specifically targets areas in the left or right atrium to eliminate areas that maintain atrial fibrillation without isolating the pulmonary veins
  Other Names: Ablation; Atrial Fibrillation; Arrhythmia; Radiofrequency Ablation; Mapping; Rotors; Pulmonary Veins; Paroxysmal Atrial Fibrillation
  Arms: FIRM Ablation

SUMMARY:
* Hypothesis: Focal Impulse and Rotor Modulation (FIRM) will substantially reduce or eliminate clinical atrial fibrillation in subjects with accepted indications for catheter ablation of paroxysmal AF, compared to standard pulmonary vein isolation.
* Summary: This is a prospective randomized study to assess the safety and effectiveness of FIRM procedures only, versus standard Pulmonary Vein Isolation (PVI) procedures for the treatment of symptomatic paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
A total of 188 subjects will be enrolled-subjects will be equally (1:1) randomized between those undergoing conventional atrial fibrillation ablation with confirmation of pulmonary vein isolation (PVI) versus those actively treated with the FIRM procedure without PVI.

ELIGIBILITY:
Inclusion Criteria:

* Reported incidence of at least two (2) documented episodes of symptomatic paroxysmal atrial fibrillation (AF) during the six months preceding trial entry (at least one episode should be documented by rhythm strip or ECG).
* Attempt of at least one Class I or III anti-arrhythmia drug with failure defined as recurrence of symptomatic AF or adverse drug effect resulting in stopping the medication (drug duration and dose will be documented).
* Left atrial size <55mm in largest dimension (typically atrial septum to carina of left pulmonary veins) as measured and image documented by preoperative imaging (CT or MRI)
* Anticoagulation therapy-Oral anticoagulation required (in the case of Warfarin, therapeutic International Normalized Ratio (INR) for at least three weeks prior to randomization) for those subjects who meet two or more of the following criteria:

  1. Age 65 years or older
  2. Diabetes
  3. Prior stroke or transient ischemic attack
  4. Congestive heart failure
  5. Hypertension with systolic>165 mm Hg
* Left Ventricular Ejection Fraction ≥ 40% (obtained within 12 months prior to the procedure)
* Sustained AF-if the patient is not experiencing spontaneous, sustained AF (>10 min uninterrupted), sustained AF may be induced by burst atrial pacing with or without isoproterenol infusion in conventional clinical fashion.

Exclusion Criteria:

* Previous catheter or surgical left atrial ablation
* Structural heart disease of clinical significance including
* Congenital heart disease where either the underlying abnormality or its correction prohibits or increases the risk of ablation
* Myocardial infarction (MI) within the past three (3) months
* Any concomitant arrhythmia or therapy that could interfere with the interpretation of the results from this study
* Atrial Septal Defect closure device; Left Atrial Appendage closure device; prosthetic mitral or tricuspid valve
* Anaphylactic allergy to contrast media
* Atrial fibrillation secondary to electrolyte imbalance

  1. thyroid disease
  2. reversible non-cardiac cause
* Poor general health that, in the opinion of the investigator, will not allow the patient to be a good study candidate (i.e. other disease processes, mental capacity, etc.)
* Reversible cause of atrial fibrillation (e.g. surgery, hyperthyroidism, pericarditis)
* Contraindication to heparin and warfarin/other new oral anticoagulants (e.g. dabigatran, rivaroxaban, apixaban [when available])
* History of pulmonary embolus within one year of enrollment
* Acute pulmonary edema
* Atrial clot/thrombus on imaging such as on a trans-esophageal echocardiogram (TEE) performed within 72 hours of the procedure if deemed appropriate by the investigator
* Any history of a cerebrovascular disease-including stroke or Transient Ischemic Attack
* Any anticipation of cardiac transplantation or other cardiac surgery within the next 365 days (12 months)
* History of documented thromboembolic event within the past one year
* Diagnosed atrial myxoma
* Significant pulmonary disease
* Acute illness or active systemic infection or sepsis
* Any history of blood clotting abnormalities or bleeding tendencies unrelated to supratherapeutic anticoagulation
* Life expectancy <365 days (12 months)
* Any intracardiac thrombus, tumor. or other abnormality that precludes safe catheter introduction or manipulation
* Continuous AF episode lasting >7 days immediately prior to the procedure without any sinus rhythm
* Patients who have previously undergone cardioversion are excluded from participation in the study unless there is documentation that cardioversion has been performed within 72 hours of episode onset
* Amiodarone use in the last 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12-23 (Actual); Study Completion 2015-12-23 (Actual)

PRIMARY OUTCOMES:
Acute Ablation Success for Paroxysmal Atrial Fibrillation | 1 week
  * the termination of spontaneous or induced atrial fibrillation by ablation at an atrial fibrillation source arrhythmia location
  * the slowing of the mean atrial fibrillation rate at least by 10% by ablation at an atrial fibrillation source arrhythmia
  * evaluate safety and effectiveness of the FIRM procedures for the treatment of paroxysmal atrial fibrillation
  * freedom from major adverse events related to the procedure within 7 days of the procedure

SECONDARY OUTCOMES:
Long Term Ablation Success for Paroxysmal Atrial Fibrillation | 1 year
  * freedom from atrial fibrillation recurrence (>30sec) from 3-12 months
  * freedom from major adverse events related to the procedure within one year of the procedure

OTHER OUTCOMES:
Quality of Life | 1 year
  EuroQOL Eq-5D scores pre-ablation will be compared to those post ablation at all points separately and together

CONTACTS AND LOCATIONS:
Overall Officials: John M Miller, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States